CLINICAL TRIAL: NCT00101387
Title: Functional Impact of PENS for 65+ Chronic Low Back Pain
Brief Title: Effects of Lumbar PENS and Exercise in Older Adults With Chronic Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Christine Crawford, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01AT000985-01A2 (NIH); R01AT000985-01A2 (NIH)
Record Dates: First submitted 2005-01-10; First posted 2005-01-11 (Estimated); Last update posted 2011-02-18 (Estimated); Status verified 2011-02

CONDITIONS: Low Back Pain
Keywords: Aged; Acupuncture
MeSH Terms: conditions — Low Back Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Lumbar PENS + exercise (Experimental): Lumbar PENS twice a week for six weeks combined with general conditioning and aerobic exercise
  Interventions: Other: Lumbar PENS + General Conditioning and Aerobic Exercise
- Lumbar PENS (Active Comparator): Lumbar PENS twice a week for 6 weeks
  Interventions: Other: Lumbar PENS
- Control PENS (Placebo Comparator): Control lumbar PENS twice a week for 6 weeks
  Interventions: Other: Control Lumbar PENS
- Control PENS + exercise (Active Comparator): Control PENS twice a week for 6 weeks along with general conditioning and aerobic exercise
  Interventions: Other: Control PENS + exercise

INTERVENTIONS:
Other: Lumbar PENS + General Conditioning and Aerobic Exercise — As above
  Arms: Lumbar PENS + exercise
Other: Lumbar PENS — As above
  Arms: Lumbar PENS
Other: Control Lumbar PENS — Identical needle placement as with PENS procedure, but only control needles stimulated for 5 minutes.
  Arms: Control PENS
Other: Control PENS + exercise — as above
  Arms: Control PENS + exercise

SUMMARY:
The purpose of this study is to determine whether a form of electrical acupuncture, called percutaneous electrical nerve stimulation (PENS), can reduce pain and disability in older adults with chronic low back pain (LBP). This study will also determine the effects of general conditioning and aerobic exercise (GCAE) on chronic LBP.

DETAILED DESCRIPTION:
Each year, a significant number of elderly individuals experience at least one episode of LBP. When LBP becomes chronic, it can lead to functional and emotional impairment, increased health care utilization, and decreased quality of life. Standard treatment for LBP typically consists of non-opioid analgesics and physical therapy; however, analgesic-associated morbidity in older adults often limits their utility. This study will determine the efficacy of PENS treatment, a neuroanatomically guided form of electroacupuncture, and exercise in reducing pain in older adults with chronic LBP.

Participants will be randomly assigned to one of four treatment groups: PENS alone, PENS placebo, PENS plus GCAE, or PENS placebo plus GCAE. The treatments will be given twice weekly for 6 weeks. Pain intensity, physical function, health care utilization, and psychosocial function will be assessed with self-report and performance-based measures. These assessments will be conducted at study start, immediately after the last treatment session, and 6 months after study completion.

ELIGIBILITY:
Inclusion Criteria:

* Low back pain for at least 3 months
* Able to walk without an assistive device (e.g., cane or walker)

Exclusion Criteria:

* Serious underlying illness causing back pain
* Nerve root compression
* History of back surgery
* Has pacemaker
* Current use of blood thinners
* Major psychiatric disorder
* Chest pains or heart problems that interfere with daily activity
* Fibromyalgia

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Actual)
Dates: Start 2003-09; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Roland and Morris questionnaire | Baseline, post-intervention, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Debra K. Weiner, MD, Principal Investigator — Pain Evaluation and Treatment Institute